CLINICAL TRIAL: NCT00316992
Title: A Study of the Safety of Ramelteon in Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: Safety of Ramelteon in Subjects With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-375-068; U1111-1115-1960 (Registry Identifier: WHO)
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Insomnia; Chronic Obstructive Pulmonary Disease; Drug Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramelteon 8 mg and Placebo (Experimental)
  Interventions: Drug: Ramelteon and Placebo

INTERVENTIONS:
Drug: Ramelteon and Placebo — Ramelteon 8 mg, tablets, orally, one night only and Ramelteon placebo-matching tablets, orally, one night only.
  Other Names: Rozerem™; TAK-375

SUMMARY:
The purpose of this study is to determine if ramelteon has respiratory depressant effects in subjects with moderate to severe chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
About 30% of the adult population report sleep disturbance and 10% meet diagnostic criteria for chronic insomnia. While 20 -25% of these individuals have primary insomnia the vast majority have an additional condition such as chronic obstructive pulmonary disease. Several studies have looked at this and have estimated that 30% to 48% of the general population is affected at some time in their life with a form of insomnia that goes on for several months, and about one third of those are described as severely affected. Daytime symptoms of insomnia include tiredness, lack of energy, difficulty concentrating and irritability. Recent epidemiologic research focusing on the quality of life has identified significant insomnia related conditions or diseases that relate to work productivity, health care utilization, and risk of depression. Insomnia is associated with diminished work output, absenteeism and greater rates of accidents.

Ramelteon, is being developed as a sleep promoting agent based on agonism of melatonin receptor subtype 1 and 2. Ramelteon is marketed in the United States as Rozerem™ for the treatment of insomnia characterized by difficulty with sleep initiation.

Sleep problems are common in patients with chronic obstructive pulmonary disease. There is evidence that traditional hypnotics can cause adverse respiratory effects in insomniac populations with respiratory disorders, and so the safety and efficacy of new hypnotic agents must be ascertained in this group of patients.

This study will examine if ramelteon has respiratory depressant effects in subjects with moderate to severe chronic obstructive pulmonary disease. Study participation is anticipated to be about 6 weeks.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Body mass index between 18 and 34, inclusive.
* Clinical history of chronic obstructive pulmonary disease and a confirmatory diagnosis based on pulmonary function tests performed at the Outpatient Screening Visit, with moderate to severe airflow limitation defined by: Moderate: forced expiratory volume in one second to forced vital capacity less than 70%; 50% less than forced expiratory volume in one second; less than 80% predicted. Severe: forced expiratory volume in one second to forced vital capacity less than 70%; forced expiratory volume in one second less than 50% predicted.
* Post-bronchodilator forced expiratory volume in one second change from baseline of less than12% and not exceeding 200 ml at the Outpatient Screening Visit.
* Oxygen saturation during wakefulness greater than 90% (both supine and sitting) as assessed by pulse oximetry at the Outpatient Screening Visit.
* Oxygen saturation during sleep of greater than or equal to 80% for at least 75% of the recording period with no more than 5 continuous minutes less than 80% and with no oxygen saturation readings less than 70% as assessed by pulse oximetry at the Inpatient Screening Visit.

Exclusion Criteria

* The health of subjects using nocturnal oxygen therapy would, in the investigator's opinion, be jeopardized by the removal of oxygen therapy during inpatient study visits.
* Electrocardiographic evidence of right ventricular hypertrophy, or evidence of right heart failure.
* Apnea hypopnea index (per hour of sleep) greater than 15 during polysomnography.
* Has had an acute clinically significant illness within two weeks or has been hospitalized within four weeks of the Outpatient Screening Visit.
* History of seizures (except childhood febrile seizures).
* History of cancer, other than basal cell carcinoma, that has not been in remission for at least five years prior to the first dose of study drug. (This criterion does not include those subjects with basal cell or Stage 1 squamous cell carcinoma of the skin.)
* History of drug addiction or drug abuse within the past 12 months, as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised.
* History of alcohol abuse within the past 12 months, as defined in
* Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised and/or regularly consumes more than 14 alcoholic drinks per week, or consumed any alcoholic drinks within six hours of any PSG visits.
* Will not refrain from use of tobacco products while in the sleep laboratory.
* Any clinically important abnormal finding, other than chronic obstructive pulmonary disease, as determined by medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Current significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic, or metabolic disease, unless currently controlled and stable with protocol-allowed medication 30 days prior to the Inpatient Screening Visit.
* Hematocrit value greater than 55% at the Outpatient Screening Visit.
* Positive hepatitis panel including anti-hepatitis A virus (only immunoglobulin M is exclusionary), hepatitis B surface antigen, or anti-hepatitis C virus.
* Alanine transaminase level of greater than three times the upper limit of normal, active liver disease, jaundice or any clinically significant abnormal laboratory findings as determined by the investigator.
* Donated more than 400 mL of blood within the 90 days preceding the beginning of the study.
* Positive urine drug screen for drugs known to alter sleep-wake function (eg, barbiturates, opiates, amphetamines, cannabinoids and alcohol) at screening, or a positive breathalyzer test for alcohol at any check-in.
* Known hypersensitivity to ramelteon or related compounds, including melatonin.
* Known hypersensitivity to albuterol or related compounds.
* Participated in any other investigational study and/or taken any investigational drug within 30 days or five half-lives prior to the first dose of single-blind study medication, whichever is longer.
* Unable to discontinue the use of hypnotics for the duration of the study.
* Has used melatonin, or other drugs or supplements known to affect sleep-wake function, within one week (or five half-lives of the drug, whichever is longer) prior to the first dose of single-blind study medication.
* Any additional condition(s) that in the Investigator's opinion would prohibit the subject from completing the study or not be in the best interest of the subject.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Within one week of single-blind medication and during the entire study.

    * Hypnotics
    * Sedating Antidepressants
    * Sedating H1 antihistamines
    * Respiratory stimulants
    * Muscle relaxants
    * The use of albuterol is acceptable during reversibility testing at the Outpatient Screening Visit.
  * Melatonin and all other drugs or supplements known to affect sleep/wake function will be prohibited within one week of the first dose of single-blind medication and during the entire study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Mean oxygen saturation during sleep for the entire night measured by pulse oximetry. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1

SECONDARY OUTCOMES:
Mean oxygen saturation calculated for each hour of the night, as measured by pulse oximetry. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Mean oxygen saturation for rapid eye movement sleep stages, as measured by pulse oximetry. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Mean oxygen saturation for non- rapid eye movement sleep stages, as measured by pulse oximetry. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Minutes for which oxygen saturation was less than 80% as measured by pulse oximetry. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Minutes for which oxygen saturation was less than 90% as measured by pulse oximetry. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Apnea-hypopnea index as determined by polysomnography. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Latency to persistent sleep as determined by polysomnography. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Total sleep time as determined by polysomnography. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Sleep efficiency as determined by polysomnography. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Wake time after persistent sleep onset as determined by polysomnography. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Number of awakenings after persistent sleep as determined by polysomnography. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Percentage of time in rapid eye movement sleep as determined by polysomnography. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Percentage of time in stage 1 sleep as determined by polysomnography. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Percentage of time in stage 2 sleep as determined by polysomnography. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Percentage of time in stage 3/4 sleep as determined by polysomnography. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Latency to rapid eye movement sleep as determined by polysomnography. | Crossover Period 1 Night 1 and Crossover Period 2 Night 1
Subjective sleep latency as determined by postsleep questionnaire. | Crossover Period 1 Morning 1 and Crossover Period 2 Morning 1
Subjective total sleep time as determined by postsleep questionnaire. | Crossover Period 1 Morning 1 and Crossover Period 2 Morning 1
Subjective Sleep Quality as determined by postsleep questionnaire. | Crossover Period 1 Morning 1 and Crossover Period 2 Morning 1
Subjective number of awakenings as determined by postsleep questionnaire. | Crossover Period 1 Morning 1 and Crossover Period 2 Morning 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda Global Research and Development
Locations (8):
- United States (8):
  - Birmingham, Alabama
  - Los Angeles, California
  - Santa Monica, California
  - Naples, Florida
  - St. Petersburg, Florida
  - Louisville, Kentucky
  - Lincoln, Nebraska
  - New York, New York

REFERENCES:
- [Result] Kryger M, Roth T, Wang-Weigand S, Zhang J. The effects of ramelteon on respiration during sleep in subjects with moderate to severe chronic obstructive pulmonary disease. Sleep Breath. 2009 Mar;13(1):79-84. doi: 10.1007/s11325-008-0196-4. Epub 2008 Jun 27. PMID 18584227
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI